CLINICAL TRIAL: NCT04129658
Title: Heart Failure in Southern Sweden - Improving the Quality of Diagnosis and Treatment Through a Educational Intervention in Primary Care
Brief Title: Heart Failure in Southern Sweden
Acronym: HISS
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: 1111
Record Dates: First submitted 2019-10-15; First posted 2019-10-17 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure，Congestive; Drug Use; Patient Care
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention: The patients are registered at PHCCs who agreed to participate into the study, the patients have provided an informed consent. The PHCCs (seventeen according to the power calculation) will receive an educational outreach visit by a cardiologist, discussing evidence-based treatment. The physician will decide afterwords if the treatment will be adjusted. Blood samples and electrocardiography will be collected before the intervention, data from the EMR will be collected before and after the intervention.
  Interventions: Behavioral: Educational outreach visit
- Control: The control group will be the rest of the patients with heart failure in Southern Sweden. Data from the regional data base on medication and heath care consumption will be collected at base line and 6 and 12 months after.

INTERVENTIONS:
Behavioral: Educational outreach visit — Two-four hours of discussion between a cardiologist and the primary care physicians at the PHCC encompassing evidence-based treatment guidelines and counseling upon specific patient cases and their diagnose and treatment for congestive heart failure.
  Groups: Intervention

SUMMARY:
The aim of the study is to optimize diagnosis and treatment for patients with heart failure in Swedish primary care. Patient with the diagnose heart failure registered in the electronic medical record (EMR) at seventeen primary health care centers (PHCCs) will be invited to to participate in the study. Blood testing and electrocardiography will be performed. Data on diagnosis and medical treatment will be collected from the EMR. An educational visit with a cardiologist will be performed at the PHCC, in order to discuss evidence-based diagnoses and treatment of heart failure. Data on drug therapy and health care consumption will be collected after six and twelve months.

DETAILED DESCRIPTION:
Background Congestive heart failure is one of the most common chronic diseases worldwide, with a prevalence of 2% of the population. With approximately 30000 affected patients, congestive heart failure is also one the most common reasons for hospital admissions in people over 65 years in southern Sweden. Heart failure means lower quality of life, a larger need for hospital care due to shortness of breath and leg swelling, risk for life threatening arrhythmia and high mortality. Several evidence-based treatment modalities have demonstrated good effect on life quality and mortality. In Sweden, there are large geographical differences in compliance to treatment guidelines. According to statistics from the National Board for Health and Welfare, in the Southern part of Sweden, Skåne, only 55% of the patients with congestive heart failure are treated with the combination of angiotensin converting enzyme inhibitors or angiotensin receptor blockers along with beta blockers. The national guidelines are recommending a target level of 65%.

The aim of this study is to assess to which extent an outreach educational program involving a cardiologist in primary care can raise the number of patients with congestive heart failure receiving evidence-based treatment, to study the cost-effectiveness of the intervention and to create a biobank for future studies in the field.

Methods The study design is prospective observational, with two patient cohorts followed over time. One cohort of patients will participate in an educational/AUDIT intervention including a cardiologist and the primary care physicians responsible for the patients. The control group will be the rest of the population in Southern Sweden, receiving usual care.

Settings Patients with a heart failure diagnosis registered in the electronic medical record (EMR) in different primary health care centers (PHCCs) will be invited to participate in the intervention group. Blood tests and electrocardiography will be performed. Blood samples for a biobank will be saved following well- regulated procedures.

Data collection Data will be collected from the EMRs in a Case Report Form (CRF). Primary outcome variable is the change in the proportion of patients receiving treatment with the combination of angiotensin converting enzyme inhibitors or angiotensin receptor blockers along with beta blockers, six months after the educational intervention.

Secondary outcome variables are the change between the groups in health care consumption and mortality as well as evidence-based treatment one year from the base line.

Data analysis The power estimation indicates that 850 patients will be required to the intervention group. Data will be analyzed with descriptive statistics and group comparison analysis for the primary outcome variable (McNemar's test and/or conditional logistic regression). Secondary outcome variables will be analyzed with group comparison for independent groups (Mann-Whitney or Student's T-test). In order to adjust for different confounders, we will use regression models. Generalized estimations equations will be used since patients are clustered within the PHCCs and can therefore not be labeled as independent.

ELIGIBILITY:
Inclusion Criteria:

* patients with ICD diagnose I50, I11.0, I42 and I43 in the electronic medical journal and who have left informed consent to participate in the study

Exclusion Criteria:

* patients with ICD diagnose I42.1, I42.2
* patients where the heart failure diagnose is set on wrong grounds according to the information in the electronic medical journal, as normal NT-proBNP or/and normal ecocardiogram.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet the inclusion criteria and left informed consent, at Swedish PHCCs that have previously agreed to participate in the study. All invited PHCCs are located in the Region of Skane, Southern Sweden.
Sampling Method: Probability Sample
Enrollment: 563 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Medication change | 6 months after inclusion
  Change in proportion of patients treated with the combination angiotensin conversion enzyme-inhibitors(ACEi) or angiotensin receptor blockers (ARB) and betablockers

SECONDARY OUTCOMES:
Change in health care consumption | One year after the intervention
  Difference between the groups in change in number of visits in hospitals or primary care
Change in mortality rate | One year after the intervention
  Difference between the groups in change in number of visits in hospitals or primary care
Change in medication | Six months after the intervention
  Difference between the groups in change of medication with mineral receptor antagonists (MRA), cardiac resynchronisation therapy (CRT), other implantable devices for treatment of heart failure (ICD) and intravenous iron for patients with iron deficiency
Change in diagnostics | Six months after the intervention
  Difference between groups in change for proportion of patients getting the diagnosis with ecocardiogram and NYHA classification

CONTACTS AND LOCATIONS:
Locations (1):
- Vårdcentralen Granen, Malmo, Sweden

REFERENCES:
- [Derived] Svensson Soderberg K, Kronestedt Lundevall L, Lindow T, O Braun O, Smith JG, Sundquist K, Milos Nymberg V. Heart failure in Southern Sweden (HISS): a cross-sectional analysis of primary care patients' characteristics and physicians' adherence to guideline-directed medical therapy. BMJ Open. 2025 Nov 4;15(11):e101178. doi: 10.1136/bmjopen-2025-101178. PMID 41248346